CLINICAL TRIAL: NCT01578096
Title: Stress Management Among Latinos With Type 2 Diabetes Mellitus
Brief Title: Stress Management Among Latinos With Type 2 Diabetes
Acronym: CALMS-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Hartford Hospital (Other); UConn Health (Other); Hispanic Health Council, Inc. (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MD005879 (NIH); R01MD005879 (NIH)
Record Dates: First submitted 2012-04-12; First posted 2012-04-16 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- Diabetes education (No Intervention): Group-based diabetes education delivered to participants through community health workers
- Diabetes education plus stress management (Experimental): Group-based diabetes education plus stress management delivered to participants through community health workers
  Interventions: Behavioral: stress management

INTERVENTIONS:
Behavioral: stress management — The study is a randomized, controlled,single-site, parallel group clinical trial comparing the effectiveness of CHW led diabetes education with CHW led diabetes education plus CHW led stress management in Latinos with Type 2 Diabetes.
  Arms: Diabetes education plus stress management

SUMMARY:
The primary aims of this study are to:

1. Tailor a diabetes stress management intervention for delivery by community health workers (CHWs) serving an urban Latino population.
2. Investigate the efficacy of the stress management intervention on glycemic control.

   Secondary aims of this study are to:
3. Investigate the efficacy of the stress management intervention on stress hormones, psychosocial functioning, and stress-glucose reactivity.

Study hypothesis:

A CHW-led group-based diabetes education model enhanced with stress management education will improve glycemic control more than CHW-led group-based diabetes education alone.

ELIGIBILITY:
Inclusion Criteria:

* Latinos age 18 or older that are ambulatory
* Spanish speaking
* Diagnosed with type 2 diabetes for at least 1 year
* Hemoglobin A1c levels greater than 7.0

Exclusion Criteria:

* Medical instability or medical treatment requiring inpatient care
* Diagnoses of bipolar disorder or thought disorder (or taking medications prescribed for either); current substance abuse or dependence disorder
* Current suicidality or history of suicide attempt
* History of psychiatric hospitalization
* Taking antidepressant medications prescribed for the treatment of depression accompanied by either a) changes to the antidepressant regimen within previous 6 weeks, or b) anticipated changes to the regimen during period of study. Such patients will be deferred and re-evaluated for eligibility after 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | Baseline
  Blood will be drawn from participants and hemoglobin A1c levels will be measured
Hemoglobin A1c | 9 weeks
  Blood will be drawn from participants and hemoglobin A1c levels will be measured
Hemoglobin A1c | 6 months
  Blood will be drawn from participants and hemoglobin A1c levels will be measured

SECONDARY OUTCOMES:
Diabetes specific distress | Baseline
  Participants will be asked questions assessing their perspective of emotional distress from living with diabetes
Diabetes specific distress | 9 weeks
  Participants will be asked questions assessing their perspective of emotional distress from living with diabetes
Diabetes specific distress | 6 months
  Participants will be asked questions assessing their perspective of emotional distress from living with diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Pérez-Escamilla, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Bermudez-Millan A, Perez-Escamilla R, Lampert R, Feinn R, Damio G, Segura-Perez S, Chhabra J, Kanc K, Wagner JA. Night Eating Among Latinos With Diabetes: Exploring Associations With Heart Rate Variability, Eating Patterns, and Sleep. J Nutr Educ Behav. 2022 May;54(5):449-454. doi: 10.1016/j.jneb.2022.02.006. PMID 35534102
- [Derived] Wagner J, Armeli S, Tennen H, Bermudez-Millan A, Wolpert H, Perez-Escamilla R. A daily study of stressors, continuously measured glucose, and diabetes symptoms in latinos with type 2 diabetes. J Behav Med. 2021 Feb;44(1):94-103. doi: 10.1007/s10865-020-00162-1. Epub 2020 Jun 3. PMID 32494976
- [Derived] Bermudez-Millan A, Wagner JA, Feinn RS, Segura-Perez S, Damio G, Chhabra J, Perez-Escamilla R. Inflammation and Stress Biomarkers Mediate the Association between Household Food Insecurity and Insulin Resistance among Latinos with Type 2 Diabetes. J Nutr. 2019 Jun 1;149(6):982-988. doi: 10.1093/jn/nxz021. PMID 31006809
- [Derived] Bermudez-Millan A, Perez-Escamilla R, Segura-Perez S, Damio G, Chhabra J, Osborn CY, Wagner J. Psychological Distress Mediates the Association between Food Insecurity and Suboptimal Sleep Quality in Latinos with Type 2 Diabetes Mellitus. J Nutr. 2016 Oct;146(10):2051-2057. doi: 10.3945/jn.116.231365. Epub 2016 Aug 3. PMID 27489004